CLINICAL TRIAL: NCT03999905
Title: Impact of Pharmacists' Training on Oral Anticoagulant Counseling: a Randomized Control Trial Using Mystery Patient Model.
Brief Title: Impact of Pharmacists' Training on Oral Anticoagulant Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, SEGUN SHOWANDE, Principal Investigator, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PharmImpact001
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Atrial Fibrillation
Keywords: Patient counseling; Mystery patient; Oral anticoagulant; Pharmacist; Warfarin; Adverse drug reaction; Nigeria; Community pharmacists
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Participants are assigned into either arm of the study randomly. Participants in the intervention arm will receive educational training after baseline assessment while participants in the control group will receive the same training after the study had been completed.
Who Masked: Care Provider, Investigator
Masking Description: Participants were randomized into the intervention and control arm through computer-generated random numbers. the randomization was done by a neutral person. The investigators and the mystery patients were unaware of the members of the intervention arm or the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Online training on Oral anticoagulant counseling.
  Interventions: Behavioral: Counseling training
- Control Arm (No Intervention): No counseling training

INTERVENTIONS:
Behavioral: Counseling training — Online training using Moodle.
  Arms: Intervention Arm

SUMMARY:
This study evaluates the impact of community pharmacists' educational training on the nature and adequacy of counseling provided to patients on warfarin, an oral anticoagulant. Half of the community pharmacists participating in the study will receive a two-week educational training on how to adequately counsel patients on warfarin while the other half of community pharmacists will receive the same training after the study. A mystery patient model will be used in this intervention study where six different trained and standardized individuals will act as patients. Each of these mystery patients will supposedly have pulmonary embolism, deep vein thrombosis, or atrial fibrillation. The mystery patient will visit each pharmacy to buy warfarin or complain about adverse drug reaction been experienced. It is expected that pharmacists will provide relevant information and counseling to these patients on the use of the medication warfarin and how to handle the adverse drug reactions.

DETAILED DESCRIPTION:
Although direct oral anticoagulants also have their limitations (such as the risk of gastrointestinal bleeding) they are not as prominent as that of warfarin but still important to consider before prescribing to patients. These limitations associated with the use of oral anticoagulants prove that there is need for special counseling of patients placed on oral anticoagulants. Counseling, as an important aspect of drug therapy management, is somewhat technical and requires a peculiar way of providing vital information on drug therapy within the shortest possible time. Pharmacists, who are key members of the healthcare team, are tasked with this role more than others and as such this area is of optimum importance.

Proper and adequate counseling on oral anticoagulants is essential for optimal use of the drug and to reduce the number of incidence of adverse drug reactions. Adequate counseling cannot be achieved without proper training. This aspect is seen to be lacking due to the suboptimal performance discovered in research among healthcare professionals including pharmacists with regards to counseling of patients on oral anticoagulant use Mystery patients in pharmacy practice research are a very reliable means of obtaining unbiased data on pharmacists with regards to counseling. This study, therefore, is aimed at providing counseling training to community pharmacists and evaluating the impact of the training on patients indirectly using the mystery patient model.

ELIGIBILITY:
Inclusion Criteria:

* Community Pharmacists with at least one-year practice experience
* Community pharmacies that stock and dispense warfarin

Exclusion Criteria:

* Community pharmacists working in order sectors

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Change in the level of oral anticoagulant counseling | Baseline and at 2-weeks post intervention training
  Level of counseling is determined by the mnemonic WARFARINISED median score. W - When to take warfarin, A - Alcohol consumption effect, R - Risk of bleeding explanation, F - Follow-up appointments, A - Aspirin and other drugs affect the action of warfarin, R - Reason for taking warfarin, I - Interactions with food and drinks, N - Notify health professional of the medication, I - International Normalised Ration measurement, S - Skipped doses, what to do, E - End of treatment, D - Dose of warfarin
  Each of the counseling points will be scored 1 point. The minimum score will be 0 point and the maximum will be 12 points.
  Higher values indicate better counseling provided by the pharmacist while lower value indicate poor counseling .

SECONDARY OUTCOMES:
Detection of adverse drug reaction due to warfarin | Baseline and 4 week post intervention training.
  Identification and counseling on detected adverse drug reaction resulting from the use of warfarin
Detection of drug interaction with warfarin | Baseline and 4 week post intervention training.
  Identification and counseling drug interaction with warfarin

CONTACTS AND LOCATIONS:
Overall Officials: Segun J Showande, Ph.D, Study Director — University of Ibadan
Locations (1):
- Community Pharmacies in Ibadan Metropolis, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data will be made available online.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available on the Mendeley database repository six months after the completion of the study.
Access Criteria: Once the data is uploaded on the Mendeley database repository, it can be accessed easily.
URL: https://data.mendeley.com/drafts/